CLINICAL TRIAL: NCT05106231
Title: Effectiveness of Pharmacy Integrated Community Care (PICC) Improving Hemoglobin A1c (HBA1C) and Knowledge in Diabetes Mellitus (DM) Education Program
Brief Title: Effectiveness of PICC Improving HBA1C and Knowledge in Diabetes Mellitus Education
Acronym: EPICCIHKDMEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Kamarudin Bin Ahmad, Chief Pharmacist, Miri Hospital Sarawak, Clinical Research Centre, Malaysia
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: NMRR-21-767-59240
Record Dates: First submitted 2021-09-28; First posted 2021-11-03 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus; Type2 Diabetes
Keywords: diabetes mellitus; Type2 diabetes; group based intervention; patient integrated community care (PICC)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study's design will be a prospective, multicenter and parallel-design single-blind randomised controlled with two treatment groups. The trial evaluates a PICC's effectiveness in improving HBA1C involving four-session structured group-based intervention (SGBI) of a two to three-hour pharmacist-led program with follow up evaluations. The control arm will have the same syllabus without SGBI.
Who Masked: Outcomes Assessor
Masking Description: For the blinding of researchers, they remain blinded towards the stage of publication. During the post-intervention follow up, the researchers still are blinded by the participants' allocation, as the Sarawak Pharmacy Service Division keeps the participant list with group allocation. None of the instruments distributed to the participants will disclose their name and group assignment to assure the blinding among researchers who do the data analyses. Only after this study's results are published, the blinding or the codes will be broken through the return of the participants' list to the principal investigator. The Sarawak Pharmacy Service Division will maintain the randomisation codes throughout the study without disclosing them to the researchers or the participants. No breaking code procedure is necessary for this study as the intervention of this study is educational and does not involve the investigation of medicinal products (IMP).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICC arm (Experimental): Participants assigned to the intervention group will attend the PICC program, which will take four-month and each session 2.5 hours.
  Interventions: Behavioral: PICC Program
- Control arm (Active Comparator): Participants assigned to the DMTAC group will receive a standard intervention of pharmacist-led education.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: PICC Program — Participants will attend the PICC program which consists of 4 sessions that involve Visualization in Participatory Programmes (VIPP) and quizzes to evaluate retention in diabetes knowledge.
  Other Names: Pharmacy Integrated Community Care
  Arms: PICC arm
Behavioral: Control — The control arm received four sessions one-on-one education program by a pharmacist. It is a Malaysian national education pharmacy-led program to instil knowledge and inculcate medication adherence.
  Other Names: DMTAC
  Arms: Control arm

SUMMARY:
The Ministry of Health Malaysia designs an education program for diabetes mellitus under the "Know Your Medicine" campaign. The Pharmacy Integrated Community Care (PICC) program hopes to improve knowledge and self-care for diabetes mellitus patients. PICC contains four modules that will provide knowledge on diabetes mellitus in an interactive, easily understandable and fun program. The investigators want to evaluate the program's effectiveness to see its relevance to Malaysian.

PICC is an education program to give knowledge on diabetes mellitus to patients. It intended to improve self-care knowledge for patients with underlying Type 2 Diabetes Mellitus conducted the whole of Malaysia. However, in Sarawak, the investigators interested in conducting it together with this is an experimental study aiming to examine PICC's effectiveness. The study is being conducted in the nine Sarawak divisions. A minimum of 94 respondents will be participating in this study. Patient profile details will be taken with strict confidentiality.

DETAILED DESCRIPTION:
Study title: Effectiveness of Pharmacy Integrated Community Care (PICC) Improving Hemoglobin A1c (HBA1C) and Knowledge in diabetes mellitus (DM) education program

Study Population: The population will be local people living in Sarawak from multiple racial backgrounds with underlying type 2 diabetes mellitus (T2DM). The investigators recruit patients with underlying T2DM mellitus who obtain medication at each district's primary Government Health Clinic.

Study Design: The study will be a prospective, multicenter and parallel-design single-blind randomised controlled with two treatment groups. The trial evaluates a PICC's effectiveness in improving HBA1C involving a four-session structured group-based intervention (SGBI) of a two to three-hour pharmacist-led program with follow-up evaluations. The control arm will be the Diabetes Mellitus Therapy Adherence Clinic (DMTAC). DMTAC is a gold standard for pharmacy-led DM education in Malaysia and an individualised-based program.

General Objective:

1. To describe and critically appraise DM education studies in Malaysia.
2. To examine the program's effectiveness versus control in improving medication adherence with underlying T2DM in the Sarawak State of Malaysia.

Specific Objectives:

1. To measure the effectiveness of PICC in improving HbA1C, fasting blood glucose and understanding
2. To investigate the sustainability of the program.

Study endpoints/outcomes:

Primary outcome: laboratory-analysed HbA1C will be the primary outcome. Secondary outcome: Investigating knowledge and understanding of DM medication management will be evaluated using the quizzes in the PICC program.

Sample Size: A previous study has shown a standard deviation of 1.5. Suppose the actual difference between the experimental and control means is 1, 36 experimental and 36 control subjects with a probability (power) of 0.8. By estimating 30% dropout or incomplete data, a minimum sample size of 94 (47 for each group).

Study Duration: 1 October to 31 January 2022.

ELIGIBILITY:
Inclusion Criteria:

1. were non-pregnant adults >18 years of age regardless of gender or ethnicity;
2. spoke and understood Bahasa Malaysia
3. had a medical record showing haemoglobin A1c test (HbA1c) level of ≥6.3% (45 mmol/mol) and fasting plasma glucose test (FPG) ≥7.0 mmol/L
4. Patients also need to be able to provide informed consent to participate in the study

Exclusion Criteria:

1. Participants were excluded if they could not answer the quizzes independently or had a hearing or vision impairment.
2. Patients unable to read, write and speak Malay, medically unstable or unable to provide informed consent will be excluded.
3. Patients who are currently attending intensive psychological treatment, hospitalised and participating in other studies will also be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
laboratory-analysed HbA1C improvement (HbA1c level below 42mmol/mol or 6.5%) | 4 months
  PICC education influencing change in HBA1C (HbA1c level below 42mmol/mol or 6.5% -CDC guideline on diabetes) using finger prick test within 4 month.

SECONDARY OUTCOMES:
Diabetes knowledge improvement (scores in percentage) | 4 months
  PICC improved diabetic knowledge scores (score above or equal to 80% up to 100% showing good knowledge)

CONTACTS AND LOCATIONS:
Overall Officials: Kamarudin Ahmad, B.Pharm, Principal Investigator — Jabatan Farmasi, Hospital Miri
Locations (9):
- Malaysia (9):
  - Klinik Kesihatan Daro, Daro, Sarawak
  - Klinik Kesihatan Kapit, Kapit, Sarawak
  - Klinik Kesihatan Jalan Masjid Kuching, Kuching, Sarawak
  - Klinik Kesihatan Bandar Miri, Miri, Sarawak
  - Klinik Kesihatan Pusa, Pusa, Sarawak
  - Klinik Kesihatan Sarikei, Sarikei, Sarawak
  - Klinik Kesihatan Siburan, Serian, Sarawak
  - Klinik Kesihatan Jalan Oya, Sibu, Sarawak
  - Klinik Kesihatan Sri Aman, Simanggang, Sarawak

IPD SHARING:
Plan to Share IPD: No
Data collection forms are not in codes. Site investigators and participants have access to individual case report forms because the information is transparent to those involved.

REFERENCES:
- [Background] Ting CY, Adruce SAZ, Hassali MA, Ting H, Lim CJ, Ting RS, Jabar AHAA, Osman NA, Shuib IS, Loo SC, Sim ST, Lim SE. Correction to: Effectiveness and sustainability of a structured group-based educational program (MEDIHEALTH) in improving medication adherence among Malay patients with underlying type 2 diabetes mellitus in Sarawak State of Malaysia: study protocol of a randomized controlled trial. Trials. 2019 May 10;20(1):267. doi: 10.1186/s13063-019-3348-x. PMID 31077233
- [Background] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Background] Soto-Greene ML, Salas-Lopez D, Sanchez J, Like RC. Antecedents to effective treatment of hypertension in Hispanic populations. Clin Cornerstone. 2004;6(3):30-6; discussion 37-8. doi: 10.1016/s1098-3597(04)80062-0. PMID 15707260
- [Derived] Ahmad K, Anchah L, Ting CY, Lim SE. Effectiveness of a pharmacist-led, community group-based education programme in enhancing diabetes management: A multicentre randomised control trial. Contemp Clin Trials Commun. 2024 Feb 24;38:101280. doi: 10.1016/j.conctc.2024.101280. eCollection 2024 Apr. PMID 38435429
- See also: The protocol is written following the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) checklist. — https://www.spirit-statement.org/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: study protocol Version 7.0 dated February 14, 2024_archive (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT05106231/Prot_SAP_ICF_003.pdf